CLINICAL TRIAL: NCT05908526
Title: The Impact of Suvorexant on Cognitive Function and Daytime Symptoms Among Community-dwelling Older Adults With Insomnia: A Placebo-controlled, Randomized Clinical Trial Using Remote Monitoring and Ecological Momentary Assessment
Brief Title: Insomnia Treatment and EMA (Ecological Momentary Assessment) Outcomes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Emerson Wickwire, Professor, Psychiatry and Medicine; Section Head, Sleep Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-00100622
Record Dates: First submitted 2023-05-11; First posted 2023-06-18 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-09

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Surveys and Questionnaires; Neuropsychological Tests; Ecological Momentary Assessment; Actigraphy; suvorexant

STUDY DESIGN:
Intervention Model Description: The study employs a two-group (suvorexant, 20mg, qhs, versus placebo) parallel design and involves a baseline assessment, 2-day low-dose run-in, and approximately 14-day active treatment phase with intensive ambulatory monitoring via wrist actigraphy and ecological momentary assessment (EMA). Outcome assessments are conducted at two weeks while participants are on study treatment or placebo and include self-report questionnaires and objective cognitive testing administered by computer.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blind, randomized, placebo-controlled, single site clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment (Experimental): Participants will start on 10mg suvorexant, po, qhs, including instructions on dosage, expectations, and potential side effects, for two nights. Following this low-dose run-in period, individuals in the treatment condition will be increased to 20mg for a 14-day active treatment period (i.e.,16 nights taking a pill). Other assessments include self-report research questionnaires and cognitive testing (completed at baseline and post-treatment), as well as EMA surveys, daily sleep diaries, and actigraphy.
  Interventions: Behavioral: Baseline surveys, Cognitive testing and EMAs; Device: Actiwatch; Drug: suvorexant (or placebo)
- Placebo (Placebo Comparator): Participants in the control condition will take placebo (no drug) pill form, po, qhs, including instructions on dosage, expectations, and potential side effects for (16 nights taking a pill). Other assessments include self-report research questionnaires and cognitive testing, daily sleep diaries, and actigraphy.
  Interventions: Behavioral: Baseline surveys, Cognitive testing and EMAs; Device: Actiwatch; Other: Placebo

INTERVENTIONS:
Behavioral: Baseline surveys, Cognitive testing and EMAs — Outcome assessments are conducted at two weeks while participants are on study treatment or placebo and include self-report questionnaires and cognitive testing administered by computer.
  Other Names: ecological momentary assessment
Device: Actiwatch — Participants will wear an actiwatch for 16 days while completing EMA surveys. It has a small sensor that tracks motion.
  Other Names: actigraphy
Drug: suvorexant (or placebo) — FDA approved which is an orexin receptor antagonist indicated for the treatment of insomnia, characterized by difficulties with sleep onset and/or sleep maintenance.
  Other Names: Belsomra
  Arms: Treatment
Other: Placebo — An inactive substance that looks like the drug or treatment being tested.
  Other Names: no drug
  Arms: Placebo

SUMMARY:
The goal of this study is to examine the impact of suvorexant, an FDA-approved insomnia medication, on daytime symptoms (as measured by the Daytime Insomnia Symptoms Scale: cognition, positive mood, negative mood, and fatigue/sleepiness) among older adults with insomnia. The primary hypothesis is that relative to placebo, suvorexant will improve sleep and daytime symptoms. The word "placebo" refers to a harmless pill with no therapeutic effect.

DETAILED DESCRIPTION:
The study will take about six to eight weeks to complete. Participants will have a home sleep apnea test (HSAT) and complete a clinical interview. Participants will also complete a baseline assessment, which will take place over one or two days (about 3 hours total).

During the study, participants will complete research questionnaires and cognitive testing at baseline and post-baseline (after treatment). Participants will also complete brief EMA surveys (sleep diary and Daytime Insomnia Symptoms Scale) via mobile device 4 times per day for approximately 16 days; each survey will take about 2 minutes or less to complete. Participants will also wear an actigraph on the non-dominant wrist. This device looks like a wristwatch and measures ambulatory movement, a validated proxy for sleep.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual - Fifth Edition (DSM-5) diagnostic criteria for insomnia disorder.
* Insomnia Severity Index total score >10.
* Insomnia symptoms must include problems with wake after sleep onset.
* Insomnia symptom duration > 6 months.
* Baseline self-reported total sleep time < 6.5 hours per night.

Exclusion Criteria:

* High risk for untreated organic sleep disorders other than insomnia (narcolepsy, periodic limb movement disorder, etc) as determined by structured clinical interview and investigator clinical judgment.
* Current diagnosis of a major untreated psychiatric disorder(s).
* History of serious suicide attempt within past 5 years.
* History of alcohol or substance abuse (including prescription medication abuse) within past 5 years.
* Heavy alcohol consumption (e.g., >5 drinks per day or > 14 drinks per week.
* Heavy caffeine use [(>2 cups of coffee/day (equivalent).
* Current tobacco or nicotine use.
* History of previous allergic reaction, sensitivity, or severe side effects to sedative hypnotics.
* CYP3A inhibitors.
* Refusal to discontinue or intention to initiate OTC or other sleep aids during study period.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emerson M Wickwire, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers at this time.

REFERENCES:
- [Background] Shiffman S, Stone AA, Hufford MR. Ecological momentary assessment. Annu Rev Clin Psychol. 2008;4:1-32. doi: 10.1146/annurev.clinpsy.3.022806.091415. PMID 18509902
- [Background] Buysse DJ, Thompson W, Scott J, Franzen PL, Germain A, Hall M, Moul DE, Nofzinger EA, Kupfer DJ. Daytime symptoms in primary insomnia: a prospective analysis using ecological momentary assessment. Sleep Med. 2007 Apr;8(3):198-208. doi: 10.1016/j.sleep.2006.10.006. Epub 2007 Mar 23. PMID 17368098
- [Background] Herring WJ, Connor KM, Snyder E, Snavely DB, Zhang Y, Hutzelmann J, Matzura-Wolfe D, Benca RM, Krystal AD, Walsh JK, Lines C, Roth T, Michelson D. Suvorexant in Elderly Patients with Insomnia: Pooled Analyses of Data from Phase III Randomized Controlled Clinical Trials. Am J Geriatr Psychiatry. 2017 Jul;25(7):791-802. doi: 10.1016/j.jagp.2017.03.004. Epub 2017 Mar 8. PMID 28427826
- [Background] Wickwire EM, Verceles AC, Chen S, Zhao Z, Rogers VE, Wilckens KA, Buysse DJ. Smart Phone/Ecological Momentary Assessment of Sleep and Daytime Symptoms Among Older Adults With Insomnia. Am J Geriatr Psychiatry. 2023 May;31(5):372-378. doi: 10.1016/j.jagp.2023.01.020. Epub 2023 Feb 1. PMID 36813640
- [Derived] Wickwire EM, Zhou J, Chen S, Wilckens KA, Steenbergh TA, Buysse DJ, Verceles AC. Smartphone-Based Real-Time Assessment of Daytime Insomnia Symptoms With Suvorexant: A Randomized Clinical Trial. JAMA Netw Open. 2026 Jan 2;9(1):e2550186. doi: 10.1001/jamanetworkopen.2025.50186. PMID 41490112

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited to the study in several ways (i.e., volunteer lists, mailings based on EPIC searches, newspaper advertisements, online and social media advertisements, public presentations, and word of mouth and study fliers). The participants were provided with study staff contact information, and the participant called. For online and social media, advertisements, and recruitment pathways, if interested the participant would complete online preliminary screening questionnaire.
Pre-assignment Details: The study participants that were confirmed eligible were randomized to drug or placebo in a 1:1 ratio by the IDS pharmacy.
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Customized [Count of Participants; unit: Participants]
  60 to 69 years old | 12 | 12 | 24
  70 to 79 years old | 8 | 8 | 16
  80-85 years old | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 12 | 13 | 25
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Daytime Insomnia Symptoms Scale (DISS)
Description: This measure assesses daytime symptoms and functional impairments in five domains: alert cognition, fatigue, sleepiness, negative mood, and positive mood. Participants will complete this survey four times per day on their smart phone for approximately 16 days. The possible score range is 0-100, with higher scores indicating greater levels of a given construct.
Time Frame: Baseline (start of study) and end of study (before day 16).
Population: Older adults with insomnia.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment: Participants randomized to suvorexant (SUV)
- Placebo: Participants randomized to placebo (PBO)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  Alert Cognition morning | 65.96 (21.66) | 70.34 (19.63)
  Alert Cognition midday | 69.22 (20.30) | 72.32 (18.45)
  Alert Cognition afternoon | 69.72 (20.35) | 71.08 (17.89)
  Alert Cognition evening | 67.54 (19.28) | 69.05 (17.09)
  Fatigue/sleepiness morning | 36.80 (25.74) | 35.83 (28.80)
  Fatigue/sleepiness midday | 35.52 (23.94) | 34.03 (27.18)
  Fatigue/sleepiness afternoon | 33.01 (24.18) | 38.72 (25.56)
  Fatigue/sleepiness evening | 38.17 (23.09) | 43.58 (26.45)
  Negative Mood morning | 27.24 (23.76) | 21.71 (22.17)
  Negative Mood midday | 26.40 (23.27) | 21.60 (21.66)
  Negative Mood afternoon | 25.35 (22.33) | 21.79 (21.66)
  Negative Mood evening | 26.09 (22.01) | 21.02 (21.74)
  Positive Mood morning | 64.42 (21.89) | 69.09 (19.34)
  Positive Mood midday | 67.23 (20.74) | 70.90 (18.04)
  Positive Mood afternoon | 67.95 (20.29) | 69.98 (18.45)
  Positive Mood evening | 66.33 (18.99) | 69.00 (16.52)

2. Primary Outcome: Change in Insomnia Severity as Assessed by Insomnia Severity Index
Description: The Insomnia Severity Index is a brief self-report instrument that measures subjective symptoms and consequences of insomnia as well as the degree of distress caused by those difficulties. Total scores range from 0 to 28, with higher scores indicating greater insomnia severity.
Time Frame: Baseline (start of study) and end of study (before day 16).
Population: Older adults with insomnia.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -9.6 (5.4) | -5.5 (6.8)

3. Secondary Outcome: Change in Sleepiness as Assessed by Epworth Sleepiness Scale
Description: The Epworth Sleepiness Scale is a brief self-report instrument that measures daytime sleepiness. Total scores range from 0 to 24, with higher scores indicating greater severity of sleepiness.
Time Frame: Baseline (start of study) and end of study (before day 16).
Population: Older adults with insomnia
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -4.2 (3.7) | -2.3 (3.6)

4. Secondary Outcome: Change in Depression as Assessed by Patient Health Questionnaire-9
Description: The Patient Health Questionnaire-9 is a brief self-report instrument that measures depressive symptoms. Total scores range from 0 to 27, with higher scores indicating greater levels of depressive symptoms.
Time Frame: Baseline (start of study) and end of study (before day 16).
Population: Older adults with insomnia.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -2.3 (3.2) | -2.2 (4.4)

5. Secondary Outcome: Change in Anxiety as Assessed by Generalized Anxiety Disorder-7
Description: The Generalized Anxiety Disorder-7 is a brief self-report instrument that measures anxiety symptoms. Total scores range from 0 to 21, with higher scores indicating greater levels of depressive symptoms.
Time Frame: Baseline (start of study) and end of study (before day 16).
Population: Older adults with insomnia.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -3.2 (4.1) | -1.6 (4.0)

6. Secondary Outcome: Change in Cognitive Performance Assessed by the PVT (Psychomotor Vigilance Test): Lapses
Description: PVT is a computer-based, chronometric test to measure reactions to specified small changes in a changing environment. Response time is scored in seconds. Response accuracy is scored numerically, with lower numbers indicating better response accuracy.
Time Frame: Baseline (start of study) and end of study (before day 16).
Population: Older adults with insomnia. Usable data was not available for ten participants (five in each treatment group).
Measure: Mean (Standard Deviation); unit: Lapses (reaction time >500 milliseconds)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 15 | 15
Lapses (reaction time >500 milliseconds) | 3.33 (6.08) | -1.13 (4.91)

7. Secondary Outcome: Change in Cognitive Performance Assessed by the PVT (Psychomotor Vigilance Test): Median Reaction Time
Description: as for outcome 6
Time Frame: Baseline (start of study) and end of study (before day 16).
Population: Older adults with insomnia. Usable data was not available for ten participants (five in each treatment group).
Measure: Median (Standard Deviation); unit: Reaction Time (milliseconds)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 15 | 15
Reaction Time (milliseconds) | 17.97 (39.9) | -10.23 (23.0)

8. Secondary Outcome: Change in Cognitive Performance Assessed by the Stroop Test: Accuracy
Description: Stroop test is a computer-based test of colors and words to measure cognitive interference. Response time is scored in seconds. Response accuracy is scored numerically, with lower numbers indicating better response accuracy.
Time Frame: Baseline (start of study) and end of study (before day 16).
Population: Older adults with insomnia. Usable data was not available for ten participants (six in the treatment group and four in the placebo group).
Measure: Mean (Standard Deviation); unit: Number of Errors
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 14 | 16
Number of Errors | -0.02 (0.19) | 0.02 (0.09)

9. Secondary Outcome: Change in Cognitive Performance Assessed by the Stroop Test: Response Time in Milliseconds
Description: Stroop test is a computer-based test of colors and words to measure cognitive interference. Response time is scored in milliseconds. Response accuracy is scored numerically, with lower numbers indicating better response accuracy.
Time Frame: Baseline (start of study) and end of study (before day 16).
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Response time in milliseconds
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 14 | 16
Response time in milliseconds | -131.3 (626.7) | -403.6 (919.5)

10. Secondary Outcome: Change in Cognitive Performance Assessed by the Task-switching: Response Time in Milliseconds
Description: Task-switching is a computer-based, chronometric test to measure response time and response accuracy. Response time is scored in milliseconds. Response accuracy is scored numerically, with lower numbers indicating better response accuracy.
Time Frame: Baseline (start of study) and end of study (before day 16).
Population: Older adults with insomnia. Usable data was not available for six participants (three in each treatment group).
Measure: Mean (Standard Deviation); unit: Response Time (milliseconds)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 17 | 17
Response Time (milliseconds) | -158.01 (535.48) | -278.42 (630.74)

11. Secondary Outcome: Change in Cognitive Performance Assessed by the Task-switching
Description: Task-switching is a computer-based, chronometric test to measure response time and response accuracy. Response time is scored in seconds. Response accuracy is scored numerically, with lower numbers indicating better response accuracy.
Time Frame: Baseline (start of study) and end of study (before day 16).
Population: Older adults with insomnia. Usable data was not available for six participants (three in each treatment group).
Measure: Mean (Standard Deviation); unit: Number of Errors
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 17 | 17
Number of Errors | 0.01 (0.14) | 0.02 (0.09)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 16 days.
Arm/Group | Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Limitations include unknown generalizability of our non-random sample of generally well-educated individuals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-16): https://cdn.clinicaltrials.gov/large-docs/26/NCT05908526/Prot_SAP_002.pdf
  • Informed Consent Form (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT05908526/ICF_001.pdf